CLINICAL TRIAL: NCT00534456
Title: Double-Blind, Placebo Controlled, Multicenter Study to Assess the Effect of Darbepoetin Alfa Treatment on Cardiac Function and Disease Specific Biomarkers in Subjects With Symptomatic Left Ventricular Systolic Dysfunction and Anemia: An Exploratory Sub-study for the RED-HF™ Trial
Brief Title: An Exploratory Sub-study for the RED-HF™ (Reduction of Events With Darbepoetin Alfa in Heart Failure) Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060172
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Anemia; Cardiovascular Disease; Congestive Heart Failure; Heart Failure; Ventricular Dysfunction
Keywords: exploratory study; anemia; pharmacogenetics testing; biomarkers; echocardiography
MeSH Terms: conditions — Anemia; Cardiovascular Diseases; Heart Failure; Ventricular Dysfunction | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Darbepoetin alfa
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo group to receive volume and dose frequency changes resembling titration dosing in the treatment group.
  Arms: Placebo
Drug: Darbepoetin alfa — Starting dose: 0.75 mcg/kg subcutaneously Q2W. Subsequent doses: Darbepoetin alfa group to receive darbepoetin alfa titrated to achieve Hb target of 13.0 g/dL, not to exceed 14.5 g/dL.
  Arms: Active

SUMMARY:
The purpose of Study 20060172 was to measure echocardiographic parameters and biomarkers in a subgroup of study subjects enrolled in Study 20050222 (the RED-HF Trial). This substudy 20060172 was terminated early due to feasibility constraints. All subjects enrolled in 20060172 were also enrolled in Study 20050222, which is ongoing. Study data will be analyzed when Study 20050222 ends, since unblinding before then would adversely affect Study 20050222.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for Study 20060172
* Randomized into Study 20050222

Exclusion Criteria:

* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, render the subject unsuitable for accurate echocardiography, may confound the study results, or may interfere significantly with the subject's participation in Study 20060172 or in Study 20050222.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To determine whether treatment of anemia with darbepoetin alfa, in patients with heart failure and anemia, results in changes in cardiac structure and function. | 12 months

SECONDARY OUTCOMES:
Explore correlations among measures of cardiac systolic and diastolic function, surrogate markers of cardiac injury and function, and clinical outcomes in heart failure subjects treated with darbepoetin alfa or placebo. | 12 months
Investigate the effect of treatment of anemia with darbepoetin alfa on novel biomarkers relevant to the pathophysiology and progression of heart failure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com